CLINICAL TRIAL: NCT02929966
Title: Effect of Palliative Care in Patients With End Stage Pulmonary Fibrosis: a Randomized Control Pilot Study
Brief Title: Palliative Care in Pulmonary Fibrosis
Acronym: PULFIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, dr. Stefano Nava, Professor of Respiratory Medicine, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 120/2016/O/Sper
Record Dates: First submitted 2016-10-08; First posted 2016-10-11 (Estimated); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Idiophatic Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard respiratory care (Placebo Comparator): The patients will receive the usual respiratory care that included both the "classical" treatments with antifibrotic drugs and oxygen therapy
  Interventions: Other: standard respiratory care
- standard respiratory care PLUS a palliative care program (Experimental): The patients will receive the usual respiratory care that included both the "classical" treatments with antifibrotic drugs and oxygen therapy PLUS a palliative care program that includes paid to assessing physical and psychosocial symptoms
  Interventions: Other: palliative care program

INTERVENTIONS:
Other: palliative care program — The program includes psychological support, spiritual care and respiratory therapist support
  Arms: standard respiratory care PLUS a palliative care program
Other: standard respiratory care — the usual standard pharmacological care plus oxygen therapy
  Arms: standard respiratory care

SUMMARY:
The investigators will examine the effect of introducing palliative in patients with end-stage idiopathic pulmonary fibrosis, refractory to the pharmacological treatment or not deemed to be treated, on patient-reported outcomes and end-of-life care. The investigators will randomly assign patients who receive either early palliative care integrated with standard respiratory care or standard respiratory care alone.

Quality of life and symptoms will assessed at baseline and at 12 weeks The primary outcome will be the change in the quality of life and symptoms at 12 months.

DETAILED DESCRIPTION:
Advanced fibrosing interstitial lung disease (ILD) is a group of often progressive and incurable conditions.

The most common form of ILD, idiopathic pulmonary fibrosis (IPF), is associated with poor survival, and high symptom burden and poor quality of life as the disease progresses.

ILD represents an increasing proportion of patients with chronic hypoxemic respiratory failure.

Despite this poor prognosis, palliative care remains underused in patients with ILD. This may be due to under-recognition of the palliative care needs and symptom burden, or unfamiliarity and discomfort with palliative therapies.

Though oncology has largely embraced earlier integration of palliative care, which has translated into improvements in end-of-life (EOL) care for patients with lung cancer,palliative and EOL care for non-malignant diseases are now gaining increased attention.

In pulmonary disease, this research has mainly focused on COPD and demonstrated a significant burden of unmet palliative care needs and lower quality of EOL care compared with patients with cancer. Similar attention is only beginning to be paid to ILD, but symptom burden and quality of EOL care in patients with ILD have yet to be quantified, and furthermore none has so far investigated the possible role of palliative care in these patients.

The investigators will examine with the present study the effect of introducing palliative in patients with end-stage idiopathic pulmonary fibrosis, refractory to the pharmacological treatment or not deemed to be treated, on patient-reported outcomes and end-of-life care. The investigators will randomly assign patients who receive either early palliative care integrated with standard respiratory care or standard respiratory care alone.

Quality of life and symptoms will assessed at baseline and at 12 weeks The primary outcome will be the change in the quality of life and symptoms at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of idiophatic pulmonary fibrosis
* resting partial arterial oxygen pressure (PaO2) < 60 mmHg
* Decline in Forced Vital Capacity (FVC) > 10% in the last 6 months
* stage 3 according to the GAP index

Exclusion Criteria:

* active treatment with antifibrotic drug
* concomitant cancer

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
clinical status and quality of life | 12 months
  Maugeri Respiratory Questionnaire reduced form
depression | 12 months
  Center for Epidemiologic Studies Depression score (C-ESDs)
dyspnea score | 12 months
  Borg scale

SECONDARY OUTCOMES:
survival | 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Sant'Orsola Malpighi Hospital, Bologna, Province
  - San'Orsola Malpighi Hospital, Bologna ITALY, Bologna

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bassi I, Guerrieri A, Carpano M, Gardini A, Prediletto I, Polastri M, Curtis JR, Nava S. Feasibility and efficacy of a multidisciplinary palliative approach in patients with advanced interstitial lung disease. A pilot randomised controlled trial. Pulmonology. 2023 Dec;29 Suppl 4:S54-S62. doi: 10.1016/j.pulmoe.2021.11.004. Epub 2021 Dec 28. PMID 34969647